CLINICAL TRIAL: NCT04893239
Title: Exploratory Study to Assess Delivery of LMN-201 Components Via Enteric Capsules in the Gut of Individuals With Ostomies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lumen Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDI01
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: C. Diff. Infections
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 LMN-201 Anti-toxin B VHH-1 (Experimental)
  Interventions: Biological: LMN-201 Anti-toxin B VHH-1
- Cohort 1 LMN-201 Anti-toxin B VHH-2 (Experimental)
  Interventions: Biological: LMN-201 Anti-toxin B VHH-2
- Cohort 1 LMN-201 Anti-toxin B VHH-3 (Experimental)
  Interventions: Biological: LMN-201 Anti-toxin B VHH-3
- Cohort 4 LMN-201 VHH 1, 2, 3 (Experimental)
  Interventions: Biological: LMN-201 Anti-toxin B VHH-1, VHH-2, VHH-3

INTERVENTIONS:
Biological: LMN-201 Anti-toxin B VHH-1 — Components of LMN-201
  Arms: Cohort 1 LMN-201 Anti-toxin B VHH-1
Biological: LMN-201 Anti-toxin B VHH-2 — Components of LMN-201
  Arms: Cohort 1 LMN-201 Anti-toxin B VHH-2
Biological: LMN-201 Anti-toxin B VHH-3 — Components of LMN-201
  Arms: Cohort 1 LMN-201 Anti-toxin B VHH-3
Biological: LMN-201 Anti-toxin B VHH-1, VHH-2, VHH-3 — Components of LMN-201
  Arms: Cohort 4 LMN-201 VHH 1, 2, 3

SUMMARY:
This is a Phase 1, single-site, open label, exploratory study to assess delivery of LMN-201 components via enteric capsules in the gut of individuals with ostomies.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the clinical trial
* Able and willing to provide informed consent
* Stable ostomy (no revisions in the last 6 months)
* At least 19 years old
* Medically stable, but may be on medications for chronic conditions

Exclusion Criteria:

* Unable or unwilling to provide adequate informed consent
* Non-English speakers
* Clinically significant disease
* Women who are pregnant, intending to become pregnant, or breastfeeding
* Use of anti-diarrheal medicine
* Suffer gastroparesis
* Opioid use

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Mason, Study Director — Lumen Bioscience, Inc.
Locations (3):
- Australia (3):
  - Wesley Medical Research Limited, Auchenflower, Queensland
  - Coastal Digestive Health, Maroochydore, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2 LMN-201 VHH 1, 2, 3: LMN-201 Anti-toxin B VHH-1, VHH-2, VHH-3: Components of LMN-201
Period: Overall Study
Arm/Group | Cohort 1 LMN-201 Anti-toxin B VHH-1 | Cohort 1 LMN-201 Anti-toxin B VHH-2 | Cohort 1 LMN-201 Anti-toxin B VHH-3 | Cohort 2 LMN-201 VHH 1, 2, 3
Started | 2 | 2 | 2 | 6
Completed | 2 | 2 | 2 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults aged 19 and above with mature ileostomy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 LMN-201 Anti-toxin B VHH-1 | Cohort 1 LMN-201 Anti-toxin B VHH-2 | Cohort 1 LMN-201 Anti-toxin B VHH-3 | Cohort 2 LMN-201 VHH 1, 2, 3 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 6 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (13.4) | 57.5 (3.5) | 57 (11.3) | 54.3 (12.1) | 56.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4 | 8
  Male | 0 | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 6 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 2 | 2 | 2 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of Capsules and/or Transit Markers in Ostomy Fluid by Visual Observation
Description: Count of participants with the presence or absence of capsules and/or transit markers at each collection timepoint in ostomy fluid by visual observation.
Time Frame: Arrival (baseline), Predose (immediately before dosing), and up to 12 hours post dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 LMN-201 Anti-toxin B VHH-1 | Cohort 1 LMN-201 Anti-toxin B VHH-2 | Cohort 1 LMN-201 Anti-toxin B VHH-3 | Cohort 2 LMN-201 VHH 1, 2, 3
Number analyzed (Participants) | 2 | 2 | 2 | 6
Participants
  Arrival (Baseline) | 0 | 0 | 0 | 0
  Pre-dose (immediately before dosing) | 0 | 0 | 0 | 0
  1 hour post-dose | 0 | 0 | 0 | 0
  2 hours post-dose | 0 | 1 | 0 | 0
  3 hours post-dose | 1 | 2 | 0 | 3
  4 hours post-dose | 1 | 2 | 1 | 4
  5 hours post-dose | 2 | 2 | 1 | 2
  6 hours post-dose | 1 | 1 | 1 | 4
  7 hours post-dose | 1 | 0 | 2 | 3
  8 hours post-dose | 1 | 0 | 1 | 3
  9 hours post-dose | 1 | 0 | 1 | 1
  10 hours post-dose | 0 | 0 | 2 | 0
  11 hours post-dose | 1 | 0 | 0 | 0
  12 hours post-dose | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 hours
Arm/Group | Cohort 1 LMN-201 Anti-toxin B VHH-1 | Cohort 1 LMN-201 Anti-toxin B VHH-2 | Cohort 1 LMN-201 Anti-toxin B VHH-3 | Cohort 4 LMN-201 VHH 1, 2, 3
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 LMN-201 Anti-toxin B VHH-1 (N=2) | Cohort 1 LMN-201 Anti-toxin B VHH-2 (N=2) | Cohort 1 LMN-201 Anti-toxin B VHH-3 (N=2) | Cohort 4 LMN-201 VHH 1, 2, 3 (N=6)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT04893239/Prot_000.pdf